CLINICAL TRIAL: NCT04332107
Title: Azithromycin for Prevention of Disease Progression in Patients With Mild or Moderate COVID-19
Brief Title: Azithromycin for COVID-19 Treatment in Outpatients Nationwide
Acronym: ACTION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Thomas M. Lietman (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Pfizer (Industry); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Thomas M. Lietman, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-30504
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin (Experimental): 1.2g of oral azithromycin
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Azithromycin — Participants will be shipped a single 1.2 g dose of oral azithromycin
  Arms: Azithromycin
Drug: Placebos — Participants will be shipped a dose of matching placebo
  Arms: Placebo

SUMMARY:
This individually randomized telemedicine-based trial aims to evaluate the efficacy of a single dose of azithromycin for prevention of progression of COVID-19 in patients with a recent positive SARS-CoV-2 test who are not currently hospitalized.

DETAILED DESCRIPTION:
Identification of a safe, effective treatment for individuals with mild or moderate COVID-19 that prevents disease progression and reduces hospitalization would reduce the burden on the health system. High dose hydroxychloroquine is being evaluated for SARS-CoV-2 prevention and COVID-19 disease treatment, but has a high risk of a number of potentially severe adverse events. Recent evidence has indicated that the broad-spectrum macrolide azithromycin may have some activity against coronaviruses. Here we propose an individually-randomized, placebo-controlled trial to determine the efficacy of a single dose of azithromycin for prevention of COVID-19.

Potential participants will undergo remote eligibility screening with study staff prior to enrollment. Upon determination of eligibility and signing electronic informed consent documents, participants will be emailed baseline study forms and will be mailed their randomized study treatment. At the end of the study (21 days), participants will be emailed a final study questionnaire. Note that there will no contact between study staff and participants in this trial, minimizing risk of infection spread.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a positive SARS-CoV-2 test and test results received within the previous seven days
* Not currently hospitalized
* Willing and able to receive study drug by mail
* Willing and able to do the study questionnaires at baseline, day 3, 7, 14, 21 days via email or over the phone
* No known allergy or other contraindication to macrolides
* Age 18 years or older at the time of enrollment
* No known history of prolongation of the QT interval (eg. History of torsades de pointes, congenital long QT syndrome, bradyarrhthmia)
* No recent use of hydroxychloroquine within the past 7 days for participants >55 years of age
* Not currently taking nelfinavir or warfarin (Coumadin)
* Provision of informed consent
* Not currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Oldenburg, ScD, MPH, Principal Investigator — University of California, San Francisco; Thuy Doan, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Oldenburg CE, Pinsky BA, Brogdon J, Chen C, Ruder K, Zhong L, Nyatigo F, Cook CA, Hinterwirth A, Lebas E, Redd T, Porco TC, Lietman TM, Arnold BF, Doan T. Effect of Oral Azithromycin vs Placebo on COVID-19 Symptoms in Outpatients With SARS-CoV-2 Infection: A Randomized Clinical Trial. JAMA. 2021 Aug 10;326(6):490-498. doi: 10.1001/jama.2021.11517. PMID 34269813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 22, 2020 and March 16, 2021, 604 participants were screened and 263 participants were enrolled. All study recruitment and enrollment was done remotely.
Pre-assignment Details: Common reasons for ineligibility included a negative COVID-19 test result (n=70), a COVID-19 test result outside of the 7 day window (n=118), could not be reached for consent (n=73), and under the age of 18 (19). A total of 341 screened participants were excluded.
Period: Day 3
Arm/Group | Azithromycin | Placebo
Started | 171 | 92
Completed | 145 | 72
Not Completed | 26 | 20
Not completed — Lost to Follow-up | 23 | 14
Not completed — Missing outcome data | 3 | 6
Period: Day 14
Arm/Group | Azithromycin | Placebo
Started | 148 (Those who had missing measurements at Day 3 but were not completely lost-to-followup were allowed to continue with the trial.) | 78 (Those who had missing measurements at Day 3 but were not completely lost-to-followup were allowed to continue with the trial.)
Completed | 131 | 70
Not Completed | 17 | 8
Not completed — Lost to Follow-up | 13 | 4
Not completed — Missing outcome data | 4 | 4
Period: Day 21
Arm/Group | Azithromycin | Placebo
Started | 135 (Those who had missing measurements at Day 14 but were not completely lost-to-followup were allowed to continue with the trial.) | 74 (Those who had missing measurements at Day 14 but were not completely lost-to-followup were allowed to continue with the trial.)
Completed | 125 | 72
Not Completed | 10 | 2
Not completed — Lost to Follow-up | 10 | 2

BASELINE CHARACTERISTICS:
Population: A single participant in the Azithromycin group did not have baseline symptom information.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 171 | 92 | 263
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [35 to 49] | 44 [35 to 51] | 43 [35 to 50]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 participants did not provide their gender information
  Participants
    number analyzed (Participants) | 168 | 92 | 260
    Female | 117 | 57 | 174
    Male | 51 | 35 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 94 | 56 | 150
  Latinx/Hispanic | 49 | 27 | 76
  Non-Hispanic Black | 11 | 1 | 12
  Non-Hispanic Asian | 6 | 3 | 9
  Mixed Race | 4 | 3 | 7
  Non-Hispanic Middle Eastern/Arab | 2 | 1 | 3
  Prefer not to answer | 1 | 0 | 1
  Not reported (missing) | 4 | 0 | 4
  Non-Hispanic Native American | 0 | 1 | 1
Geographic region [Count of Participants; unit: Participants]
  West | 79 | 40 | 119
  Southeast | 38 | 14 | 52
  Southwest | 24 | 16 | 40
  Midwest | 21 | 16 | 37
  Northeast | 9 | 6 | 15
Alcohol consumption >3x/week [Count of Participants; unit: Participants] | 23 | 9 | 32
Current cigarette smoker [Count of Participants; unit: Participants] | 13 | 5 | 18
Current marijuana user [Count of Participants; unit: Participants] | 9 | 6 | 15
Current e-cigarette/vaping [Count of Participants; unit: Participants] | 8 | 2 | 10
Current cigar use [Count of Participants; unit: Participants] | 1 | 1 | 2
Comorbidities [Count of Participants; unit: Participants]
  Asthma | 21 | 11 | 32
  Hypertension | 20 | 12 | 32
  Diabetes | 5 | 5 | 10
  Chronic obstructive pulmonary disease | 4 | 0 | 4
  Chronic kidney disease | 1 | 1 | 2
  Cancer | 1 | 0 | 1
  Stroke | 1 | 1 | 2
Recent macrolide use (<30 days) [Count of Participants; unit: Participants] | 22 | 11 | 33
Recent hydroxychloroquine use (<7 days) [Count of Participants; unit: Participants] | 1 | 0 | 1
Current medications [Count of Participants; unit: Participants]
  ACE/ARB inhibitor | 15 | 14 | 29
  Metformin | 4 | 3 | 7
  Omeprazole | 1 | 1 | 2
  Tacrolimus | 1 | 0 | 1
Current vitamin/supplement use [Count of Participants; unit: Participants]
  Vitamin D | 64 | 37 | 101
  Vitamin C | 61 | 33 | 94
  Multivitamin | 52 | 27 | 79
  Zinc | 49 | 20 | 69
  Omega-3 fatty acid | 14 | 6 | 20
Self-reported symptoms [Count of Participants; unit: Participants]
  Multiple symptoms | 152 | 82 | 234
  Cough | 111 | 61 | 172
  Fatigue | 107 | 55 | 162
  Fever | 87 | 40 | 127
  Myalgia | 82 | 40 | 122
  Anosmia | 80 | 39 | 119
  Sore throat | 71 | 37 | 108
  Diarrhea | 45 | 20 | 65
  Shortness of breath | 45 | 17 | 62
  Dizziness | 39 | 15 | 54
  Abdominal pain | 29 | 12 | 41
  None | 12 | 6 | 18
  Conjunctivitis | 8 | 2 | 10
Number of symptoms [Median (Inter-Quartile Range); unit: Number of symptoms] | 5 [3 to 6] | 4 [3 to 6] | 4 [3 to 6]
Duration of symptoms prior to test [Median (Inter-Quartile Range); unit: days] | 3 [2 to 4.5] | 3 [2 to 4] | 3 [2 to 4]
Days between positive test and enrollment [Median (Inter-Quartile Range); unit: days] | 3 [1 to 5] | 2 [1 to 4] | 3 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Symptom Free at Day 14
Description: Binary assessment of whether the participant is experiencing any symptoms at Day 14 (yes or no)
Time Frame: 14 days
Population: Percentage of participants who were symptom free at day 14 by randomized treatment group, overall and in pre-specified subgroups. Note that a single participant in the Azithromycin group did not have baseline symptom information.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 131 | 70
Participants
  Overall | 66 | 35
  Age <= 60 years: number analyzed (Participants) | 121 | 62
  Age <= 60 years | 61 | 31
  Age > 60 years: number analyzed (Participants) | 10 | 8
  Age > 60 years | 5 | 4
  Asymptomatic at baseline: number analyzed (Participants) | 10 | 4
  Asymptomatic at baseline | 9 | 3
  Symptomatic at baseline: number analyzed (Participants) | 120 | 66
  Symptomatic at baseline | 57 | 32

2. Secondary Outcome: Viral Load - Nasal Swab
Description: Viral load by self-collected nasal swab
Time Frame: 3 days
Population: Participants whose samples were received back by the study team. The trial was terminated for futility, funding was withdraw and samples not analyzed and will never be analyzed
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Viral Load - Saliva Swab
Description: Viral load by self-collected saliva swab
Time Frame: 3 days
Population: Participants whose samples were received back by the study team. The trial was terminated for futility, funding was withdraw and samples not analyzed and won't ever be analyzed
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mortality
Description: All-cause mortality
Time Frame: 14 days
Population: This outcome is based on the 125 participants in the azithromycin group and the 72 participants in the placebo group who completed the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 125 | 72
Participants | 0 | 0

5. Secondary Outcome: Adverse Events
Description: Percentage of participants experiencing adverse events, including gastrointestinal side effects and rash
Time Frame: 3 days
Population: Adverse events were recorded at day 3 of the trial via an online questionnaire. Other adverse events were recorded in an open text field and included stomach cramps, light headedness, fatigue, ansomia, cough, and painful respiration.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 145 | 72
Participants
  Diarrhea | 60 | 12
  Nausea | 32 | 7
  Abdominal Pain | 25 | 1
  Vomiting | 5 | 2
  Rash | 4 | 2
  Other | 10 | 3
  None | 9 | 45

6. Secondary Outcome: Positive SARS-CoV-2 Test - Nasal Swab
Description: Prevalence of positive SARS-CoV-2 test by self-collected nasal swab
Time Frame: 3 days
Population: as for outcome 3
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Positive SARS-CoV-2 Test - Saliva Swab
Description: Prevalence of positive SARS-CoV-2 test by self-collected saliva swab
Time Frame: 3 days
Population: as for outcome 3
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Positive SARS-CoV-2 Test - Rectal Swab
Description: Prevalence of positive SARS-CoV-2 test by self-collected rectal swab
Time Frame: 3 days
Population: as for outcome 3
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Genetic Macrolide Resistance Determinants
Description: Prevalence of genetic macrolide resistance determinants by self-collected rectal swab
Time Frame: 3 days
Population: as for outcome 3
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Secondary Outcomes Through Day 21
Description: Prevalence of cough, fever, myalgia, anosmia, shortness of breath, fatigue, conjunctivitis, and orthostatic symptoms through Day 21
Time Frame: Cumulative over 21 days reported (assessed at 3, 7, 14, 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 125 | 72
Participants
  Absence of symptoms | 71 | 43
  Fever | 1 | 1
  Cough | 14 | 13
  Diarrhea | 4 | 1
  Abdominal pain | 0 | 1
  Anosmia | 12 | 9
  Conjunctivitis | 2 | 0
  Sore throat | 4 | 4
  Shortness of breath | 16 | 4
  Myalgia | 5 | 3
  Fatigue | 32 | 17
  Dizziness | 6 | 3
  Other | 10 | 9

11. Secondary Outcome: Number of Participants With Emergency Room Visits
Description: Number of emergency room visits <24 hours
Time Frame: 21 days
Population: Number of patients who reported emergency room visit information through Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 125 | 72
Participants | 18 | 2

12. Secondary Outcome: Number of Household Members With COVID-19 (Confirmed or Symptomatic)
Description: Number of household members with confirmed or symptomatic COVID-19 through Day 21
Time Frame: 21 days
Population: Includes the total number of participants from 69 households in the placebo group and 134 households in the azithromycin group
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 522 | 278
Participants | 33 | 20

13. Secondary Outcome: Number of Participants That Died
Description: Deaths within the study
Time Frame: 21 days
Population: Participants that completed the day 21 questionnaire were included in this secondary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 125 | 72
Participants | 0 | 0

14. Secondary Outcome: Number of Participants Reporting Hospitalization
Description: Number of hospitalizations defined as a hospital stay or ER stay longer than 24 hours through 21 days post enrollment
Time Frame: 21 Days
Population: Number of patients who reported hospitalization information through Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 125 | 72
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: 21 days
Description: Participants completed a survey at day 3 where they were asked if they had experienced any of the following symptoms since they took their study medication to assess possible adverse events: vomiting, nausea, diarrhea, rash, or abdominal pain. Participants were asked at every time point if they had stayed in a hospital setting (defined as in the emergency department or admitted to the hospital for >= 24 hours) and/or if they had visited an emergency department or urgent care center.
Arm/Group | Azithromycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/72
Other Adverse Events (participants affected / at risk) | 132/145 | 25/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=145) | Placebo (N=72)
Diarrhea (Gastrointestinal disorders) | 60 | 12
Nausea (Gastrointestinal disorders) | 32 | 7
Abdominal pain (Gastrointestinal disorders) | 25 | 1
Vomiting (Gastrointestinal disorders) | 5 | 2
Other (Gastrointestinal disorders) | 10 | 3

LIMITATIONS AND CAVEATS:
This trial was terminated early by the DSMC for futility on March 16, 2021. Therefore, we were not able to complete the analysis for all secondary outcomes because funds were returned to the sponsor following the completion of the study.

Please note that the number of participants varies by period as participants could opt to complete some questionnaires but not others. For example, a participant may skip the day 3 questionnaire, but complete the day 14 questionnaire.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT04332107/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT04332107/SAP_001.pdf